CLINICAL TRIAL: NCT04999150
Title: A Split-Mouth Randomized Clinical Trial for the Comparison of Corticotomy and Micro-Osteoperforations During Canine Retraction: A Pilot Study
Brief Title: Comparison of Corticotomy and Micro-Osteoperforation During Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Collaborators: University of Zagreb (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPR MSC IRB B0710118
Record Dates: First submitted 2021-08-09; First posted 2021-08-10 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Malocclusion, Class I/II
Keywords: Corticotomy; MOP; Tooth movement
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: a split-mouth randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Each patient was randomly assigned an identification number (S1-S13) by picking a sealed envelope. The randomization of IDs to the right or left side for MOP was accomplished with a 1:1 allocation ratio, using a computer-generated research randomizer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Corticotomy (Active Comparator): 1. A full-thickness labial mucoperiosteal flap was reflected.
  2. Two vertical corticotomies (1 mesial and 1 distal to the canine) were performed . The cortical bone was cut 2 to 3 mm below the alveolar crest towards the apex until bone marrow was exposed.
  3. Cortical-cancellous bone grafts (0.5cc; PuraGraft, Kingwood, TX) were placed at the corticotomy sites.
  4. The mini-screws were placed.
  5. A nickel-titanium (NiTi) closed-coil spring was placed and secured with a 0.014"SS ligature wire at the canine and mini-screw. A Dontrix gauge (Orthopli Corp., Philadelphia, PA) was used to measure the force (150g).
  Interventions: Procedure: Corticotomy
- Micro-Osteoperforation (Experimental): 1. MOPs were performed with a stainless-steel manual drill tip that had 1.6mm diameter with an adjustable depth set to 5mm (Excellerator® RT; Propel Orthodontics, Milpitas, CA).
  2. Six perforations were made along 2 parallel vertical lines (each line with 3 holes spaced ~2mm apart) distal to the canine and perpendicular to the buccal cortical bone.
  3. The mini-screws were placed.
  4. A NiTi closed-coil spring was placed and secured with a 0.014"SS ligature wire at the canine and mini-screw. A Dontrix gauge was used to measure the force (150g).
  Interventions: Procedure: Micro-Osteoperforations

INTERVENTIONS:
Procedure: Micro-Osteoperforations — MOPs were performed with a stainless-steel manual drill tip that had 1.6mm diameter with an adjustable depth set to 5mm (Excellerator® RT; Propel Orthodontics, Milpitas, CA).
  Six perforations were made along 2 parallel vertical lines (each line with 3 holes spaced ~2mm apart) distal to the canine and perpendicular to the buccal cortical bone.
  The mini-screws were placed. A NiTi closed-coil spring was placed and secured with a 0.014"SS ligature wire at the canine and mini-screw. A Dontrix gauge was used to measure the force (150g)
  Other Names: MOP
  Arms: Micro-Osteoperforation
Procedure: Corticotomy — A full-thickness labial mucoperiosteal flap was reflected. Two vertical corticotomies (1 mesial and 1 distal to the canine) were performed. The cortical bone was cut 2 to 3 mm below the alveolar crest towards the apex, until bone marrow was exposed.
  Cortical-cancellous bone grafts (0.5cc; PuraGraft, Kingwood, TX) were placed at the corticotomy sites.
  The mini-screws were placed. A nickel-titanium (NiTi) closed-coil spring was placed and secured with a 0.014"SS ligature wire at the canine and mini-screw. A Dontrix gauge (Orthopli Corp., Philadelphia, PA) was used to measure the force (150g)
  Arms: Corticotomy

SUMMARY:
Corticotomy and micro-osteoperforation (MOP) have been proven to accelerate tooth movement and shorten orthodontic treatment time, compared to conventional treatment. MOP is less invasive; however, it is unclear whether it is as effective as a corticotomy. The purpose of this study was to compare the maxillary canine retraction achieved by these techniques.

DETAILED DESCRIPTION:
Thirteen patients (5 females, 8 males; mean age, 18.07±6.74 years) with healthy permanent dentition requiring the extraction of maxillary first premolars were included in a split-mouth randomized clinical trial. Subjects with previous orthodontic or endodontic treatment of canines were excluded. At least 3 months post-extraction, MOPs, and corticotomies were performed distal to the canines. Mini-screws with closed-coil springs (150g) were used for canine retraction. Dental casts were attained at baseline (T0) and 3 months post-intervention (T1). Calibrated examiners measured the distances from the canine to the second premolar on both sides. A Signed-rank sum test was used to compare canine retraction achieved in 3 months (T0-T1) in two sides

ELIGIBILITY:
Inclusion Criteria:

* Healthy permanent dentition requiring the extraction of maxillary first premolars with less than 8mm of maxillary anterior crowding

Exclusion Criteria:

* Previous orthodontic or endodontic treatment of the canines

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2020-09-26 (Actual)

PRIMARY OUTCOMES:
Canine retraction | 3 months
  Amount of tooth movement (in mm) attained by the maxillary canines after retracting them

CONTACTS AND LOCATIONS:
Overall Officials: Augusto R Elias, DMD,MSD, Study Director — Assitant Dean of Research
Locations (1):
- UPR Medical Sciences Campus, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Jacox LA, Little SH, Ko CC. Orthodontic tooth movement: The biology and clinical implications. Kaohsiung J Med Sci. 2018 Apr;34(4):207-214. doi: 10.1016/j.kjms.2018.01.007. Epub 2018 Feb 3. PMID 29655409
- [Background] Aboul-Ela SM, El-Beialy AR, El-Sayed KM, Selim EM, El-Mangoury NH, Mostafa YA. Miniscrew implant-supported maxillary canine retraction with and without corticotomy-facilitated orthodontics. Am J Orthod Dentofacial Orthop. 2011 Feb;139(2):252-9. doi: 10.1016/j.ajodo.2009.04.028. PMID 21300255
- [Background] Frost HM. The regional acceleratory phenomenon: a review. Henry Ford Hosp Med J. 1983;31(1):3-9. No abstract available. PMID 6345475
- [Background] Verna C. Regional Acceleratory Phenomenon. Front Oral Biol. 2016;18:28-35. doi: 10.1159/000351897. Epub 2015 Nov 24. PMID 26599115
- [Background] Aboalnaga AA, Salah Fayed MM, El-Ashmawi NA, Soliman SA. Effect of micro-osteoperforation on the rate of canine retraction: a split-mouth randomized controlled trial. Prog Orthod. 2019 Jun 3;20(1):21. doi: 10.1186/s40510-019-0274-0. PMID 31155698
- [Background] Cheung T, Park J, Lee D, Kim C, Olson J, Javadi S, Lawson G, McCabe J, Moon W, Ting K, Hong C. Ability of mini-implant-facilitated micro-osteoperforations to accelerate tooth movement in rats. Am J Orthod Dentofacial Orthop. 2016 Dec;150(6):958-967. doi: 10.1016/j.ajodo.2016.04.030. PMID 27894545
- [Background] Fischer TJ. Orthodontic treatment acceleration with corticotomy-assisted exposure of palatally impacted canines. Angle Orthod. 2007 May;77(3):417-20. doi: 10.2319/0003-3219(2007)077[0417:OTAWCE]2.0.CO;2. PMID 17465647
- [Background] Leethanakul C, Kanokkulchai S, Pongpanich S, Leepong N, Charoemratrote C. Interseptal bone reduction on the rate of maxillary canine retraction. Angle Orthod. 2014 Sep;84(5):839-45. doi: 10.2319/100613-737.1. Epub 2014 Mar 4. PMID 24592904
- [Background] Alikhani M, Raptis M, Zoldan B, Sangsuwon C, Lee YB, Alyami B, Corpodian C, Barrera LM, Alansari S, Khoo E, Teixeira C. Effect of micro-osteoperforations on the rate of tooth movement. Am J Orthod Dentofacial Orthop. 2013 Nov;144(5):639-48. doi: 10.1016/j.ajodo.2013.06.017. PMID 24182579
- [Background] AMLER MH, JOHNSON PL, SALMAN I. Histological and histochemical investigation of human alveolar socket healing in undisturbed extraction wounds. J Am Dent Assoc. 1960 Jul;61:32-44. doi: 10.14219/jada.archive.1960.0152. No abstract available. PMID 13793201
- [Background] Arreghini A, Lombardo L, Mollica F, Siciliani G. Torque expression capacity of 0.018 and 0.022 bracket slots by changing archwire material and cross section. Prog Orthod. 2014 Sep 25;15(1):53. doi: 10.1186/s40510-014-0053-x. PMID 25329505
- [Background] Pandis N, Walsh T, Polychronopoulou A, Katsaros C, Eliades T. Split-mouth designs in orthodontics: an overview with applications to orthodontic clinical trials. Eur J Orthod. 2013 Dec;35(6):783-9. doi: 10.1093/ejo/cjs108. Epub 2013 Feb 1. PMID 23376899
- [Background] Alikhani M, Alansari S, Sangsuwon C, et al. Micro-osteoperforations: Minimally invasive accelerated tooth movement. Semin Orthod. 2015; 21(3): 162-169.
- Available data/document: Study Protocol: B0710118 — https://irbrcm.rcm.upr.edu/